CLINICAL TRIAL: NCT05380856
Title: Sacral Neuromodulation for Patients With Multiple Sclerosis With Neurogenic Lower Urinary Tract, Bowel and Sexual Dysfunction. A Multicenter Double-blind, Placebo-controlled Randomized Clinical Trial.
Brief Title: Sacral Neuromodulation for Neurogenic Lower Urinary Tract, Bowel and Sexual Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Copenhagen (Other); Université de Nantes (Other); University of Ostrava (Other)
Responsible Party: Principal Investigator, Hanne Kobberø, Principal investigator, MD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OdenseOUH
Record Dates: First submitted 2021-12-22; First posted 2022-05-19 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Neurogenic Dysfunction of the Urinary Bladder; Multiple Sclerosis; Sacral Neuromodulation; Bowel Dysfunction; Sexual Dysfunction; Quality of Life
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Multiple Sclerosis; Intestinal Diseases; Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: After the implantation of the IPG the patients will be grouped into three strata:
  1. Patients with urgency frequency syndrome and/or urgency incontinence: at least 50% decrease in number of voids and/or number of leakages and/or increased voided volume and/or more than 50% reduction in pad weight
  2. Patients with chronic urinary retention: at least 50% decrease in post void residual and/or reduction in number of CISC
  3. Patients with a combination of urgency frequency syndrome and/or urgency incontinence and chronic urinary retention: at least 50% decrease in number of voids and/or number of leakages and/or more than 50% reduction in pad weight, and/or at least 50% decrease in post void residual and/or a reduction in number of CISC
  After four months all IPG´s are turned on.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: After a month of optimization where the IPG is turned on at subsensory stimulation the participants will be randomly assigned to either intervention or placebo group with a 1:1 allocation as per a computer generated randomization schedule by a clinician who is not involved in the assessment of the clinical outcome.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- IPG turned ON (Active Comparator): Continous neuromodulation
  Interventions: Device: Turning ON the neuromodulator
- IPG turned OFF (Placebo Comparator): No neuromodulation
  Interventions: Device: Turning OFF the neuromodulator

INTERVENTIONS:
Device: Turning ON the neuromodulator — IPG on
  Other Names: INTERSTIM X SYSTEM
  Arms: IPG turned ON
Device: Turning OFF the neuromodulator — IPG OFF
  Other Names: INTERSTIM X SYSTEM
  Arms: IPG turned OFF

SUMMARY:
A multi-center double-blinded placebo-controlled randomized clinical trial.

The patients will be randomized into two groups.

To investigate the efficacy of SNM to improve the key bladder diary variables compared to placebo (i.e. sham) for patients with MS having refractory neurogenic lower urinary tract dysfunction (NLUTD).

After first step SNM-procedure and a 3-4 weeks test period patients with more than 50% improvement in the key bladder diary variables will have the IPG implanted. After a month of optimization patients will into two groups: IPG ON or IPG OFF.

Period of randomization: four months. Number anticipated to be included: 60 patients

DETAILED DESCRIPTION:
Patients with MS often suffer from pelvic-organ dysfunctions, i.e. lower urinary tract (LUT), bowel and sexual dysfunction, aside their cerebral affection. Sacral neuromodulation (SNM) is a reversible minimal invasive procedure affecting the function of the aforementioned pelvic organs. Changes in bladder, bowel and sexual function will be monitored.

Primary outcome:

Success of SNM for lower urinary tract dysfunction as improvement of at least 50% in the key bladder diary variables (i.e. number of voids and/or number of leakages, post void residual) compared to the baseline values.

Secondary outcome:

To assess the changes in bladder, bowel and sexual function due to SNM by using subjective patient reported outcome measures, quality of life and global assessment score,

* To assess the changes in urodynamic variables,
* To assess the safety of SNM for NLUTD and
* To register the implantation characteristics and the need for reprogramming

Data will be collected at Baseline 1: At inclusion Baseline 2: At evaluation after a three weeks test period Baseline 3: At randomization Baseline 4: At the end of study

The time frame of the RCT is six months

Patients with improvements of bowel symptoms only will be excluded from the trial but followed with the same questionnaires for the same time.

The patients will be followed-up every 6 months for a total of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Refractory neurogenic lower urinary tract dysfunction (nLUTD) defined by visual analogue scale on treatment satisfaction ranging from 0 to 100 (100 means maximal satisfaction with the current treatment). All patients indicating satisfaction less than 50 are considered non-responders/having refractory overactive bladder (OAB) to current treatment
* No effect of medical treatment defined by antimuscarinics, beta3-agonist and alpha-blocker.
* Patients having refractory nLUTD who intend to try SNM for relief of their symptoms
* Expanded Disability Status Scale (EDSS) < 5 and no progression of neurological disease within 6 months
* Written informed consent
* Able to understand the information given about the project

Exclusion Criteria:

* EDSS > 5, neurological disease with severe progression within the last 6 months and/or unable to manage the electronic devices
* Age < 18 years
* Any other urological pathology but nLUTD
* Bladder Pain Syndrome/Interstitial cystitis
* Any other intestinal or gynecological pathology but neurological conditional symptoms
* Current pelvic malignancy or clinically significant pelvic mass
* Previous pelvis radiotherapy
* Bladder injections with botulinum neurotoxin type A within 6 months before inclusion in trial
* Unable to manage the electronic devices
* Inability to give an informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Success of SNM for neurogenic lower urinary tract dysfunction | Six months
  Success is defined as improvement of at least 50% in the key bladder diary variables, i.e. number of voids and/or number of leakages, post void residual volumen, compared to the baseline values using BLADDER DIARY for three days before inclusion and at evaluation.
Male bladder function | Six months
  Male lower urinary tract symptoms (MLUTS) by standard International Consultation on Incontinence Questionnaire (ICIQ)-MLUTS 10/06.
  Scale ranges from 0 to 44 points. Higher score indicate greater impact of individual symptoms for the patient.
  Changes will be compared to basal data.
Female bladder function | Six months
  Female lower urinary tract symptoms (FLUTS) by standard questionnaire ICIQ-FLUTS 12/07.
  Scale ranges from 0 to 48 points. Higher score indicate greater impact of individual symptoms for the patient.
  Changes will be compared to basal data.

SECONDARY OUTCOMES:
Changes in bladder volume | Six months
  Change in bladder volume measured in ml before and after implantation of implantable pulse generator for sacral neuromodulation
Changes in bladder sensation Mangler | Six months
  Changes in bladder sensation measured in ml before and after implantation of implantable pulse generator for sacral neuromodulation
Bowel function | Eight months
  Bowel function by standard questionnaire ICIQ-B (04/08). Scale ranges from 0 to 75 points. Higher score indicate greater impact of individual symptoms for the patient.
  Changes will be compared to basal data.
Male sexual function | Six months
  Male sexual function by standard questionnaire (07/05). Scale ranges from 0 to 12 points. Higher score indicate greater impact of individual symptoms for the patient.
  Changes will be compared to basal data.
Female sexual function | Six months
  Female sexual function by standard questionnaire (09/05). Scale ranges from 0 to 14 points. Higher score indicate greater impact of individual symptoms for the patient.
  Changes will be compared to basal data.
Quality of life by standard questionnaire EQ-5D-5L | Six months
  The EQ-5D-5L is a standard measure of health-related quality of life. EQ-5D-5L consists of two components: a health state profile and a visual analog scale (VAS). EQ-5D health state profile comprises 5 dimensions:
  mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems.
  The 5D-5L systems are converted into a single index utility score between 0 to 1, where a higher score indicates a better health state.
  The VAS records the participant's health on a 0-100 mm VAS scale, with 0 indicating "the worst health you can imagine" and 100 indicating "the best health you can imagine". Higher scores of EQ VAS indicate better health

OTHER OUTCOMES:
Adverse events | Six months
  Rate of adverse events evaluated by the Medical Device Coordination Group, (MDCG)-202010/1, safety reporting in clinical investigations of medical devices under the Regulation (EU) 2017/745
Global assessment scale | Six months
  5 point Likert scale evaluated by: Very satisfied - satisfied - neutral - unsatisfied - very unsatisfied
Implantation Characteristics | Six months
  The lowest stimulation value in mA will be monitored and number of the re-programming

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Kobberø, Principal Investigator — Odense University Hospital; Mads H Poulsen, Study Director — Odense University Hospital; Morten Blaabjerg, Study Chair — Odense University Hospital; Helle H Nielsen, Study Chair — Odense University Hospital; Mikkel Fode, Study Chair — Herlev/Gentofte
Locations (1):
- Odense University Hospital, Odense, Fyn, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The study plan will be uploaded online at the Data Management Plan (DMP) Online of the University of Southern Denmark. See website below.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From 2027 and for ten years
Access Criteria: Log in to DMP is required.
URL: https://dmponline.deic.dk/plans

REFERENCES:
- [Derived] Kobbero H, Krhut J, Zvara P, Pedersen TB, Fode M, Nielsen HH, Poulsen MH. Sacral Neuromodulation for Neurogenic Lower Urinary Tract, Bowel and Sexual Dysfunction in Patients With Multiple Sclerosis: A Pilot Trial. Neurourol Urodyn. 2025 Jun;44(5):1109-1119. doi: 10.1002/nau.70052. Epub 2025 Apr 14. PMID 40223778